CLINICAL TRIAL: NCT05319340
Title: Optimization of Anticoagulant Therapy in Outpatient Practice
Brief Title: I.M. Sechenov First Moscow State Medical University (Sechenov University)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 678657
Record Dates: First submitted 2021-03-03; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-03

CONDITIONS: Anticoagulants
Keywords: Rivaroxaban Dabigatran Apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anticoagulants arm (Other): The study embraces patients who are advised to take the anticoagulant therapy (as per the European Society of Cardiology Guidelines). The study evaluates the compliance with the anticoagulant therapy, safety and effectiveness, mortality
  Interventions: Other: prescribing anticoagulant therapy

INTERVENTIONS:
Other: prescribing anticoagulant therapy — Patients who need anticoagulants were consulted by a cardiologist with subsequent recommendations

SUMMARY:
Single-institution uncontrolled open-label trial.

DETAILED DESCRIPTION:
The single-institution uncontrolled open-label trial is to optimize the anticoagulant therapy in the out-patient practice.

The study embraces patients who are advised to take the anticoagulant therapy for some reasons. The study has two phases - a retrospective part and a concurrent part. At the first phase, researchers analyze the compliance with the anticoagulant therapy in the real clinical practice. At the concurrent phase, researchers conduct a single-institution uncontrolled open-label trial to evaluate the effectiveness, safety of the anticoagulant therapy and compliance with it at the antithrombotic therapy control ward, and estimate the glomerular filtration rate in patients taking the anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* the age above 18
* indications for the anticoagulant therapy
* informed consent for inclusion into trials

Exclusion Criteria:

* denial to proceed in the trial

Non-inclusion criteria:

pregnancy and lactation

* Intracerebral hemorrhage within three preceding months
* severe mental disorders* which could possibly affect the anticoagulant therapy dosage schedule
* anemia and a decrease in Hb by ˂100 GM/DL*
* active gastroduodenal ulcer
* active bleeding during the preceding month
* other intensive bleeding instances as per the TIMI Score within three weeks before the inclusion
* severe hepatic impairment for over 10 points under the Child-Pugh Score
* oncology disease with the life expectancy less than one year

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-01-15; Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
kidney compliance with the anticoagulant therapy and its safety and trends in the kidney function | Evaluation of GFR, bleeding and thrombotic complications after 2 years
  During a visit to the clinic, the patient will be surveyed and tested for the creatinine level
death due to any cause | in six years after the anticoagulant therapy is prescribed
  phone survey when patients are invited to the clinic
cardiovascular mortality | Evaluation of GFR, bleeding and thrombotic complications and cardiac mortality after 2 years
  Phone survey when patients are invited to the clinic. The term cardiovascular mortality means a set of fatal heart attacks, fatal strokes, sudden death, fatal thromboembolism.
kidney function trend | Evaluation of GFR, bleeding and thrombotic complications and cardiac mortality after 3 years
  phone survey when patients are invited to the clinic for testing the creatinine level and further estimation of the glomerular filtration rate
intensive bleeding | Evaluation of GFR, bleeding and thrombotic complications and cardiac mortality after 6 years
  phone survey when patients are invited to the clinic.

SECONDARY OUTCOMES:
frequency of thromboembolic events | in 1-2-3-6 years after the anticoagulant therapy is prescribed
  patients will be surveyed upon their visit to the clinic. Thromboembolic events shall mean non-fatal embolic strokes, systemic embolism, acute coronary syndrome (to be corroborated with documents).

OTHER OUTCOMES:
minor bleeding | in 1-2-3-6 years after the anticoagulant therapy is prescribed
  Minor bleeding shall mean any visually observed bleeding, including that discovered with various imaging methods, which cause a decrease in HB by less than 30 GM/DL or Ht by less than 9%.

CONTACTS AND LOCATIONS:
Overall Officials: Zukhra Salpagarova, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)

IPD SHARING:
Plan to Share IPD: No
ethics committee requirement

REFERENCES:
- [Background] Chashkina MI, Kozlovskaya NL, Andreev DA, Ananicheva NA, Bykova AA, Salpagarova ZK, Syrkin AL. [Prevalence of Advanced Chronic Kidney Disease in Patients with Nonvalvular Atrial Fibrillation Hospitalized in Cardiology Departments]. Kardiologiia. 2020 Mar 5;60(2):41-46. doi: 10.18087/cardio.2020.2.n823. Russian. PMID 32345197